CLINICAL TRIAL: NCT05376735
Title: An Exploratory Randomised Control Trial of a Single Session Intervention Combined With In-situ Socially Assistive Robot to Promote Emotion Regulation Competence in University Students
Brief Title: Randomised Control Trial of an Intervention to Promote Emotion Regulation Strategies in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); Stony Brook University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR/DP-21/22-28406
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Emotion Regulation
Keywords: emotion regulation; in-situ intervention; university students
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purrble intervention + Single Session Intervention (Experimental): The Purrble intervention takes the form of an interactive plush toy, designed to be handed over to the child and support in-the-moment soothing.
  When the Purrble is picked up, it emits a frantic heartbeat that slows down if the person uses calm stroking movements. If the Purrble is soothed for long enough, it transitions into a purring vibration indicating a calm, content state.
  The Single Session Intervention has been co-produced with university students and clinical experts (Prof Jessica Schleider), combining the theories of emotion regulation with the qualitative experiences of students in open trial.
  The result follows a traditional SSI structure (cf., Schleider et al 2020), including
  1. Initial guided reflection exercise
  2. Short interactive psychoeducation
  3. Personalised action plan
  The SSI will be accessible by students on a website and be both desktop and mobile browser friendly. The full process should not take students longer than 30 minutes.
  Interventions: Behavioral: Purrble intervention; Behavioral: Single Session Intervention
- Treatment as usual / Waiting list (No Intervention): Participants in the control group will be given a Purrble & access to the online SSI intervention before the academic term ends, after 4 week follow-up questionnaires are completed.

INTERVENTIONS:
Behavioral: Purrble intervention — The intervention takes the form of an interactive plush toy, designed to be handed over to the child and support in-the-moment soothing.
  The Purrble is introduced to the student as an anxious creature that may need kind attention from humans. When picked up, the Purrble emits a frantic heartbeat that slows down if the child uses calm stroking movements. If it's soothed for long enough, it transitions into a purring vibration indicating a calm, content state.
  Logic model underlying the intervention:
  Level 1: in-the-moment soothing support to students in emotional moments when they would attempt to practice emotion regulation (ER) strategies to calm down.
  Level 2: mechanisms that facilitate long-term engagement with the intervention, building on positive subjective experience of Level 1.
  Level 3: shift in students' ER practices and implicit beliefs about emotion, after repeated experience of Levels 1-2.
  Arms: Purrble intervention + Single Session Intervention
Behavioral: Single Session Intervention — The SSI has been co-produced with university students and clinical experts, combining the theories of ER with the qualitative experiences of students in open trial.
  The result follows a traditional SSI structure (cf., Schleider et al 2020), including
  * Initial guided reflection exercise (helping understand one's experience with Purrble in the 1st week).
  * Short interactive psychoeducation, introducing the concept of window of tolerance, the Process Model of Emotions (Gross2015), and specific ways in which Purrble can help students down-regulate emotions within the context of the process model.
  * Action plan to identify: moments when Purrble could be useful, what ER strategies they would like to use in those moments, what obstacles they may encounter, and how to overcome them.
  The SSI will be accessible by students on a website and be both desktop and mobile browser friendly. The full process should not take students longer than 30 minutes.
  Other Names: SSI
  Arms: Purrble intervention + Single Session Intervention

SUMMARY:
The primary aim of the proposed Randomised Control study is to investigate the effects of a socially assisted robot (i.e. Purrble) and a bespoke Single Session Intervention (SSI) on students' anxiety (measured by GAD7) over the period of the academic term (in comparison to a wait-listed student group).

Secondary aims include investigating the effects of the Purrble and SSI on students' depression, emotion regulation processes, and quantitative and qualitative (interviews) measures of engagement with the intervention.

DETAILED DESCRIPTION:
Need among college students for accessible mental health support is high: for example, the WHO World Mental Health International College Student project,(Auerbach et al., 2018) involving 13,984 first-year college students from eight countries, found that 31% of the respondents screened positive for depression, anxiety, or alcohol use disorder. Yet, access to professional support has long remained low, with waitlists for counseling on many campuses being weeks to months long (cf., for example Brown 2018). Digital technologies, including apps, have been proposed as one possible means of 'filling in the gaps' in extant mental health care support for college students - but most apps suffer from low usability in real-world settings (Torous et al, 2018), are not equipped to serve in-the-moment coping needs (e.g., they involve user-initiated psychoeducation modules rather than opportunities to practice and grow skills when they are needed most) and often show high drop-out rates (Musiat et al, 2014).

There thus is a clear need to harness digital technologies to create usable, engaging, evidence-supported mental health supports that may be used flexibly based on when students need them most (e.g. when stress levels are particularly high and coping skills most warrant deployment); ideally also as an adjunct completing existing counselling service.

In the pilot work last year (n=80, open trial at Oxford) the investigators evaluated one such possible tool-Purrble-designed to provide a student-centred, in-the-moment emotion regulation support. Study goals centred on testing usability/usage patterns during 8-week in-situ deployment, perceived usefulness over the same period, and links between use and symptoms in high-anxiety university students (GAD-7 > 10 at sign-up). The results have been promising, with large effects sizes on GAD7 scores over the period of the term (d~0.9), the majority of students perceived the Purrble intervention as useful with 61% reporting in the last survey that it helped their mental health, and detailed a range of positive outcomes in qualitative interviews (e.g., it helped them calm down and ground themselves in the present moment when they are feeling anxious, stressed or lonely, or be more gentle and kind with themselves -rather than harsh and judgmental- when feeling overwhelmed).

However, the open trial pilot study did not include a control or waitlisted group and thus more rigorous investigation of these promising effects is needed - leading to the current study.

ELIGIBILITY:
Inclusion Criteria:

* Currently registered as a student at Oxford University (under- or postgraduate) at the time of the study
* Currently living in the UK at the time of the study
* Aged 18-25
* GAD7 score >= 10 (Löwe, 2008)
* Consistent internet and computer/laptop/smartphone access
* Able to read and write in English

Exclusion Criteria:

* Not an Oxford University student currently living in the UK at the time of the study
* Not within age range
* GAD7 score < 10 (Löwe, 2008)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2022-07-17 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
Anxiety (measured by GAD7) -- pre/mid/post | Three times during the 4-week long deployment period: pre, mid and post deployment
  The primary aim is to investigate the effects of Purrble + SSI intervention on students' changes in anxiety over the period of academic term (in comparison to a wait-listed student group).
  Overall changes in anxiety throughout the deployment will be measured by the Generalised Anxiety Disorder Assessment (GAD-7), a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder. Each item asks the individual to rate the severity of their symptoms over the past two weeks (Splitzer et al 2006).
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions.
  Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Anxiety (measured by GAD2) -- weekly | Once a week for the 4-week long deployment period
  The primary aim is to investigate the effects of Purrble + SSI intervention on students' changes in anxiety over the period of academic term (in comparison to a wait-listed student group).
  Weekly changes in anxiety will be measured with the Generalized Anxiety Disorder 2-item (GAD-2): a very brief and easy to perform initial screening tool for generalized anxiety disorder. Each item asks the individual to rate the severity of their symptoms over the past two weeks (Kroenke et al 2007). A score of 3 points is the preferred cut-off for identifying possible cases and in which further diagnostic evaluation for generalized anxiety disorder is warranted. Using a cut-off of 3 the GAD-2 has a sensitivity of 86% and specificity of 83% for diagnosis generalized anxiety disorder.

SECONDARY OUTCOMES:
Depression -- pre/mid/post | Three times during the 4-week long deployment period: pre, mid and post deployment
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' depression over the period of academic term (in comparison to a wait-listed student group).
  Measured by the PHQ-9: a depression module which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. The maximum score is 27 (9 questions x maximum 3 points per question). Depression severity is graded based on the PHQ-9 score:
  * None 0-4
  * Mild 5-9
  * Moderately 10-14
  * Moderately severe 15-19
  * Severe 20-27
Depression -- weekly | Once a week for the 4-week long deployment period
  We will also track changes in depression on the PHQ-2 (Kroenke et al, 2003) on a weekly basis. This module uses a subset of the PHQ-9 questions ("Little interest or pleasure in doing things", "Feeling down, depressed or hopeless") on the same scoring scale ("0" (not at all) to "3" (nearly every day)).
Emotion regulation (beliefs ) -- pre/mid/post | Three times during the 4-week long deployment period: pre, mid and post deployment
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' emotion regulation processes over the period of academic term (in comparison to a wait-listed student group).
  Student-reported beliefs about emotion regulation will be measured by ER beliefs 'questionnaire (Ford et al 2018). Specifically, students will answer 4 questions on a five point likert scale (strongly disagree --> strongly agree): "If I want to, I can change the emotions that I have."; "I can learn to control my feelings."; "No matter how hard I try, I can't really change the emotions that I have."; "The truth is, I have very little control over my emotions."
Emotion regulation (self-efficacy) -- pre/mid/post | Three times during the 4-week long deployment period: pre, mid and post deployment
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' emotion regulation processes over the period of academic term (in comparison to a wait-listed student group).
  Student-reported capability of regulating / managing own emotion will be measured by the self-efficacy version of the Emotion Regulation Questionnaire (ERQ-SE; Goldin 2012).
Engagement with the Purrble intervention - open ended | Once a week for the 4-week long deployment period
  A secondary aim includes investigating the engagements with the Purrble + SSI intervention over the period of academic term.
  Measured by a bespoke survey informed by the pilot study (Dauden Roquet et al 2022). The questions inquire about Purrble use and perceived usefulness. Items are rated on a 0 to 4 scale unless otherwise specified.
  1. How often did participants engage with Purrble this week? If not at all, why do participants think that was?
  2. On average, did engaging with Purrble make any difference to how participants felt at the time?
  3. In what contexts has Purrble been most useful to participants? <open-ended>
     Have there been any situations in which Purrble has been useful to participants? <open-ended>
  4. Have there been any situations participants hoped Purrble could help with, but it didn't really work? <open-ended>
  In what contexts has Purrble been least useful to participants? <open-ended>
Engagement with the Purrble intervention - TWEETS | week 2 and week 4 of the active deployment phase
  A secondary aim includes investigating the engagements with the Purrble + SSI intervention over the period of academic term .
  Measured by an adapted version of Twente Engagement with eHealth Technologies Scale (TWEETS; Kelders et al 2020)
Engagement with the Single Session Intervention | Once after completing the online SSI programme (week 1)
  Measured by a program feedback scale (adapted for this study). Items rated on a 0 (really disagree) to 4 (really agree) scale unless otherwise specified.
  1. I enjoyed the program
  2. I understood the program
  3. This program was easy to use
  4. I tried my hardest during the program
  5. I think the program would be helpful to other university students
  6. I would recommend this program to a friend going through a hard time
  7. I agree with the program's message
  8. What did participants like about the program? Please share as many true thoughts and feelings as participants would like << open-ended, text area >>
  9. What would participants change about the program? Please share as many true thoughts and feelings as participants would like << open-ended, text area >>
Hopefulness -- weekly | Once a week for the 4-week long deployment period
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' depression over the period of academic term (in comparison to a wait-listed student group).
  Measured by:
  --> The State Hope Scale (Snyder et al, 1996) is a 6-item self-report measure of ongoing goal-directed thinking (agency and pathways). Responses are rated on an 8-point Likert scale ranging from 1 (Definitely True) to 8 (Definitely False) with higher scores indicative of greater state hopefulness.
Hopelesness -- weekly | Once a week for the 4-week long deployment period
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' depression over the period of academic term (in comparison to a wait-listed student group).
  Measured by:
  --> The Beck Hopelessness Scale (Beck, 1988) provides a self-report measure of one's negative expectations regarding the future. It consists of 20 true-false items arrayed within three factors: Feelings about the future, loss of motivation, and future expectations. The total score is a sum of item responses. Scores ranging from: 0 to 3 within the normal range, 4 to 8 mild hopelessness, 9 to 14 moderate hopelessness, and scores greater than 14 identify severe hopelessness.
Emotion regulation -- weekly | Once a week for the 4-week long deployment period
  A secondary aim includes investigating the effects of Purrble + SSI intervention on changes in students' emotion regulation processes over the period of academic term (in comparison to a wait-listed student group).
  We will administer weekly a single item anchoring item measuring the perceived change in their ability to cope with emotions 'this week'. Item is rated on a 0 (much less able) to 4 (a lot more able) scale unless otherwise specified: Since participants' last survey (one week ago), how much have participants felt able to cope with their emotions?

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auerbach RP, Mortier P, Bruffaerts R, Alonso J, Benjet C, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Murray E, Nock MK, Pinder-Amaker S, Sampson NA, Stein DJ, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. J Abnorm Psychol. 2018 Oct;127(7):623-638. doi: 10.1037/abn0000362. Epub 2018 Sep 13. PMID 30211576
- [Background] Torous J, Nicholas J, Larsen ME, Firth J, Christensen H. Clinical review of user engagement with mental health smartphone apps: evidence, theory and improvements. Evid Based Ment Health. 2018 Aug;21(3):116-119. doi: 10.1136/eb-2018-102891. Epub 2018 Jun 5. PMID 29871870
- [Background] Brown JSL. Student mental health: some answers and more questions. J Ment Health. 2018 Jun;27(3):193-196. doi: 10.1080/09638237.2018.1470319. Epub 2018 May 16. No abstract available. PMID 29768071
- [Background] Musiat P, Goldstone P, Tarrier N. Understanding the acceptability of e-mental health--attitudes and expectations towards computerised self-help treatments for mental health problems. BMC Psychiatry. 2014 Apr 11;14:109. doi: 10.1186/1471-244X-14-109. PMID 24725765
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Goldin PR, Ziv M, Jazaieri H, Werner K, Kraemer H, Heimberg RG, Gross JJ. Cognitive reappraisal self-efficacy mediates the effects of individual cognitive-behavioral therapy for social anxiety disorder. J Consult Clin Psychol. 2012 Dec;80(6):1034-40. doi: 10.1037/a0028555. Epub 2012 May 14. PMID 22582765
- [Background] Ford BQ, Lwi SJ, Gentzler AL, Hankin B, Mauss IB. The cost of believing emotions are uncontrollable: Youths' beliefs about emotion predict emotion regulation and depressive symptoms. J Exp Psychol Gen. 2018 Aug;147(8):1170-1190. doi: 10.1037/xge0000396. Epub 2018 Apr 5. PMID 29620380
- [Background] Kelders SM, Kip H, Greeff J. Psychometric Evaluation of the TWente Engagement with Ehealth Technologies Scale (TWEETS): Evaluation Study. J Med Internet Res. 2020 Oct 9;22(10):e17757. doi: 10.2196/17757. PMID 33021487

DOCUMENTS (1):
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT05376735/ICF_000.pdf